CLINICAL TRIAL: NCT00959400
Title: Efficacy and Safety Study of Fentanyl Transdermal (Fentanest®)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Eduardo Pagani, CRISTÁLIA PRODUTOS QUÍMICOS FARMACÊUTICOS LTDA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT059
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pain; Palliative Care
Keywords: Fentanyl Transdermal; Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms

ARMS (1):
- Fentanyl Transdermal (Experimental)
  Interventions: Drug: Fentanyl Transdermal

INTERVENTIONS:
Drug: Fentanyl Transdermal — Fentanest® 25 mcg/h. Each patch delivers 25 mcg of fentanyl per hour continuously for 72 hours. Therefore paches must be changed every 3 days.

SUMMARY:
Eligible patients who agree to participate will migrate from oral opioids to transdermal patches and be followed for four weeks. Oral morphine will be provided as pain rescue medication. The patients will inform the adverse events and rescue medication consumption. The number of Fentanest® patches will be adjusted every visit aiming to reduce the rescue medication consumption and adverse events to a minimum. The WHO-QOL- bref (quality of life questionary) will be filled before and after the use of Fentanest®. Patients showing benefit are eligible to a 3 weeks compassionate study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged from 18 to 70 years with cancer chronic pain who received in the last 4 weeks at least 40 mg of oral morphine or equianalgesic dose of other opioids. If using adjuvant analgesics, these must be in stable doses in the last 4 weeks.

Exclusion Criteria:

* Life expectancy bellow 4 months;
* Karnofsky score < 60;
* Hypersensitivity to opioids or patches;
* Acute pain;
* Non cancer pain;
* Increased intracranial pressure;
* Conditions that prevent the patient to understand the study directions and/or give his consent;
* Neuromuscular disorders with increased risk of respiratory depression;
* Impossibility to receive rescue oral morphine; active infections;
* Fever;
* Pregnancy and nursing;
* Uncontrolled diabetes mellitus or arterial hypertension;
* Need of anticoagulation;
* Need to operate machines or vehicles;
* Important skin disorders;
* History of severe allergic reactions;
* BMI ≥ 35;
* Safety exams outrange;
* Participation in another clinical trial within the last 2 months;
* Investigator´s opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary: formulation tolerability (assessed by adverse events incidence). Co primary: formulation analgesic efficacy (assessed by rescue medication demand). | 4 weeks folow-up

SECONDARY OUTCOMES:
Establish the correspondence between the dose of oral opioids available in Brazil and number of patches required. Establish directions for secure and effective migration from oral opioids to this formulation. Quality of life improvement (WHO-QOL-bref). | 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Hospital Universitario da Universidade Federal do Maranhao, São Luís, Maranhão
  - Instituto Nacional de Cancer - Hospital do Cancer I, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade Estadual Paulista "Julio de Mesquita Filho" - Campus de Botucatu - Unesp, Botucatu, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo - HCFMUSP, São Paulo, São Paulo